CLINICAL TRIAL: NCT07269769
Title: A Phase III , Randomized, Double-blind, Placebo-Controlled, Ranibizumab Injection Loading, Multicenter Clinical Trial Comparing the Efficacy and Safety of Sanhuang Jingshiming Pills in Subjects With nAMD
Brief Title: A Clinical Trial Evaluating the Efficacy and Safety of Sanhuang Jingshiming Pills in the Treatment of nAMD
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Tasly Pharmaceutical Group Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TSL-TCM-SHJSMW-Ⅲ
Record Dates: First submitted 2025-11-25; First posted 2025-12-08 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-11

CONDITIONS: AMD
MeSH Terms: interventions — Ranibizumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental): Sanhuang Jingshiming Pills，1 sachet/dose, bid
  Interventions: Drug: Sanhuang Jingshiming/Pills placebo
- Placebo Group (Placebo Comparator): Placebo，1 sachet/dose, bid
  Interventions: Drug: Sanhuang Jingshiming/Pills placebo

INTERVENTIONS:
Drug: Sanhuang Jingshiming/Pills placebo — Ranibizumab: 1 dose/study eye (Screening/Baseline), then PRN injections
  Other Names: Ranibizumab

SUMMARY:
The purpose of the TSL-TCM-SHJSMW-Ⅲ study is to study the efficacy and safety of Sanhuang Jingshiming Pills in subjects with Neovascular Age-Related Macular Degeneration.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 50 to 85 years old (inclusive of 50 and 85 years old)
2. Meets the Western medical diagnostic criteria for neovascular age-related macular degeneration
3. Meets the TCM syndrome differentiation criteria for Qi-Yin Deficiency with Phlegm-Blood Stasis Intermingling Syndrome
4. The study eye is diagnosed with nAMD and the disease is in the active phase
5. BCVA of the study eye assessed by the ETDRS visual acuity chart ranges from 25 to 78 letters
6. Voluntarily participates in the clinical trial, signs the ICF, and is able to understand and comply with the trial procedures

Exclusion Criteria:

1. The study eye is complicated with pathologic myopia, high myopia, or secondary MNV caused by other definite diseases, glaucoma, diabetic retinopathy , retinal artery/vein occlusion , optic neuropathy (optic neuritis, optic atrophy, papilledema), macular hole, acute phase of intraocular inflammation, or other ocular diseases
2. Patients with pure PED in the study eye
3. Patients with subfoveal structural destruction or subfoveal fibrosis/scars/RPE tear/GA in the study eye
4. Patients whose FP of the study eye shows a total macular lesion area > 9 disc areas (total lesion area is defined as the sum of the areas of MNV, atrophy, scars, and fibrosis); or patients whose FP of the study eye shows a maximum macular hemorrhage area > 4 disc areas
5. Patients with CRT ≥ 700 μm in the study eye as assessed by OCT
6. Patients with opaque refractive media (e.g., vitreous hemorrhage, cataract) in the study eye precluding adequate visualization of the fundus, or with a history of vitrectomy
7. Patients planning to undergo any intraocular surgery on the study eye during the trial period
8. Patients who received pharmacologic treatment for nAMD within 2 weeks prior to randomization
9. Patients who received intravitreal anti-vascular endothelial growth factor therapy on the study eye within 4 months prior to randomization
10. Patients who received photodynamic therapy , laser photocoagulation, macular surgery, transpupillary thermotherapy , or corticosteroid therapy on the study eye within 6 months prior to randomization
11. Patients who underwent any intraocular or periocular surgery (excluding eyelid surgery) on the study eye within 3 months prior to randomization
12. Uncontrolled hypertension (systolic blood pressure ≥ 160 mmHg or diastolic blood pressure ≥ 100 mmHg while on regular antihypertensive medication)
13. History of major cardiovascular or cerebrovascular diseases, including but not limited to: ① history of myocardial infarction (MI), coronary angioplasty or bypass surgery, valvular heart disease or valvular repair, clinically significant and treatment-requiring arrhythmia, unstable angina, transient ischemic attack (TIA), cerebrovascular accident (CVA), etc., within 6 months prior to randomization; ② congestive heart failure (CHF) with New York Heart Association (NYHA) classification of Grade Ⅲ or Ⅳ
14. Laboratory test abnormalities as follows: ① platelet count ≤ 100 × 10⁹/L; ② International Normalized Ratio (INR) ≥ 1.5; ③ total bilirubin (TBIL) > 2 × upper limit of normal (ULN); ④ alanine aminotransferase (ALT) or aspartate aminotransferase (AST) > 2.5 × ULN; ⑤ serum creatinine (Scr) > 1.5 × ULN
15. Patients with severe and unstable diseases of the mental, neurological, respiratory, digestive, renal, metabolic, immune, hematologic, or other systems, as well as malignant tumors, who are assessed by the investigator as unsuitable for participation in this clinical trial
16. Presence of any contraindications listed in the package insert of ranibizumab injection (Lucentis®) or other anti-VEGF injections
17. Suspected allergy to any study drug
18. Pregnant or lactating females; males or females who plan to conceive within 30 days from signing the ICF to the end of the trial, or who cannot use effective contraceptive measures
19. Participation in another interventional clinical trial within 3 months prior to randomization
20. Other reasons deemed unsuitable for participation in this clinical trial by the investigator

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 450 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2031-12-31 (Estimated); Study Completion 2031-12-31 (Estimated)

PRIMARY OUTCOMES:
Proportion of participants with ranibizumab injections | 24 weeks

SECONDARY OUTCOMES:
Mean number of ranibizumab injections | 24 weeks
Mean days between second ranibizumab injection and baseline | 24 weeks
Change in BCVA from baseline | 24 weeks
Proportion of participants with BCVA decrease ≥5/≥10/≥15 letters | 24 weeks
Change in lesion site thickness | 24 weeks
Change in CRT from baseline | 24 weeks
Proportion of participants with new macular hemorrhage | 24 weeks
Change in maximum macular hemorrhage area | 24 weeks
Change in NEI VFQ-25 score from baseline | 24 weeks
  The Visual Function Questionnaire 25（NEI VFQ-25） has a maximum score of 100 and a minimum score of 0. The higher the score, the better vision.
Change in TCM syndrome score from baseline | 24 weeks
  There are a total of 5 projects in Traditional Chinese Medicine syndrome scale. The scale has a maximum score of 15 and a minimum score of 0. The higher the score, the more severe the disease.
Change in individual TCM syndrome score items from baseline | 24 weeks
  There are a total of 5 projects in Traditional Chinese Medicine syndrome scale. which 2 primary symptoms scored from 0 to 6 points，and 3 secondary symptoms scored from 0 to 1 point. The higher the score, the more severe the disease.
Proportion of participants by TCM syndrome efficacy | 24 weeks
  (clinical cure/marked effect/effective/ineffective）

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No